CLINICAL TRIAL: NCT03270904
Title: The Use of Moleculight i:X™ in the Management of Diabetic Foot Ulcers: A Pilot Study
Brief Title: Moleculight i:X™ in Wound Healing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VS17/99990
Record Dates: First submitted 2017-08-31; First posted 2017-09-01 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Ulcer Foot
MeSH Terms: conditions — Foot Ulcer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Interventional Treatment (Experimental): Participants in this group have been randomised to receive application of violet blue light administered by the hand held Microlight i:X device in addition to routine care of their foot ulcer. This intervention will be administered four times during the study.
  Interventions: Device: Moleculight i:X™ fluorescence imaging
- Group 2 - Usual care (No Intervention): This group receive routine care and no additional intervention.

INTERVENTIONS:
Device: Moleculight i:X™ fluorescence imaging — Moleculight i:X™ is a hand held device that emits violet blue light. By controlling distance from the wound and ambient light, Moleculight i:X™ identifies bacteria above a pre-determined concentration by identifying natural fluorescence in the bacteria cell wall.
  Arms: Group 1 - Interventional Treatment

SUMMARY:
Diabetic foot disease is a global health problem. Diabetes affects over 450million people worldwide, expected to rise to 1 in 10 people by 2040. 60-70% will lose sensation in their feet and up to 25% will develop a diabetic foot ulcer (DFU - a wound on the foot). More than half of DFUs become infected requiring hospitalisation and 20% of infections result in amputations contributing to 80% of non-traumatic amputations performed in the developed world. DFUs cost the NHS £1billion in financial year 2014-15.

A diabetic foot ulcer is a form of chronic wound. Chronic wounds are wounds that fail to progress through the normal phases of wound healing in an orderly and timely manner and become hard to heal. Almost all chronic wounds are known to have bacteria within and this is termed colonisation. Wounds can progress from being colonised to becoming infected. The concentration of bacteria can predict delayed healing or infection.

This study aims to use a novel hand held device, Moleculight i:X™, in a pilot study to investigate the clinical effectiveness and decision making associated with its use in the assessment of DFUs. Moleculight i:X™ is a hand held device that emits violet blue light. By controlling distance from the wound and ambient light, Moleculight i:X™ identifies bacteria above a pre-determined concentration by identifying natural fluorescence in the bacteria cell wall.

Patients attending a specialist DFU clinic will be screened and if eligible and consenting will be recruited. Patients will be randomised into two groups; those who receive treatments as usual (TAU) alone (in line with NICE guidelines) and those that receive TAU plus Moleculight i:X™ imaging. The main objective is to describe the proportion per group with healed DFUs at 12week follow up in these two comparable groups of 30 patients each.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years
2. Diagnosis of Diabetes (according to WHO criteria)
3. Has ulceration of the foot below the malleoli
4. Expected to comply with the treatment strategies and follow up schedule
5. Consent to foot and wound photography
6. Consent to participate (written/witnessed verbal consent)

Exclusion Criteria:

1. Has any current clinically infected diabetic foot ulcer (as per IDSA guidelines).
2. Estimated glomerular filtration rate (eGFR) <20mL/min/1.73m2 (measurements taken within 3 months of randomisation can be used if no change in intervention or vascular events have occurred)
3. Has ABPI <0.5 or opening toe pressure <30mmHg (measured within 3 months of randomisation)
4. Planned or previous treatment with corticosteroids to an equivalent dose of Prednisolone >10mg per day or other immunosuppressive therapy within 4 weeks prior to randomisation
5. Has evidence of connective tissue disorders (e.g. vasculitis or rheumatoid arthritis) and has planned or is under active treatment.
6. Has evidence of dermatological disorders (e.g. pyoderma gangrenosum or epidermolysis bullosa)
7. Has previously been randomised to the Moleculight i:X™ study
8. Lacks mental capacity and is unable to provide informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of diabetic foot ulcers healed at 12 weeks post randomisation | 12 weeks
  The proportion of diabetic foot ulcers which have healed in both group 1 and group 2 at 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rahma S, Woods J, Brown S, Nixon J, Russell D. The Use of Point-of-Care Bacterial Autofluorescence Imaging in the Management of Diabetic Foot Ulcers: A Pilot Randomized Controlled Trial. Diabetes Care. 2022 Jul 7;45(7):1601-1609. doi: 10.2337/dc21-2218. PMID 35796769